CLINICAL TRIAL: NCT06044883
Title: Role of Shear Wave Elastography in Assessment of Penile Cavernosal Elasticity and Response to Treatment by Botox Injection in Patients With Erectile Dysfunction.
Brief Title: Radiological Evaluation of the Penis Before and After a Botox Injection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Wael Ragab, Lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-191-2023
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men suffering from erectile dysfunction not responsive to phosphodiesterase-5 inhibitors (PDEI5Is) (Experimental): Our study involves male participants aged 18-70 years old suffering from erectile dysfunction and not responding to oral PDE5Is All patients are sexually active. They had no history of pelvic or spinal surgeries or trauma. Patients will be recruited from the Andrology department and outpatient clinics - Kasr Alainy- Cairo University hospitals.
  The study will be conducted in the ultrasound unit in the Radiology department- Kasr Alainy- Cairo University hospitals.
  Interventions: Procedure: Injection of Botulinum neurotoxin (BoNT); Diagnostic Test: Penile duplex and shear wave elastosonography (SWE).

INTERVENTIONS:
Procedure: Injection of Botulinum neurotoxin (BoNT) — Botulinum neurotoxin (BoNT) is produced by Clostridium botulinum, an anaerobic ,gram-positive bacterium. Poisoning with BoNT can cause botulism, resulting in generalized paralysis, respiratory failure, and death .There are seven serotypes of BoNT: A, B, C1, D, E, F, and G. BoNT-A is the most commonly used serotype for medical purposes.
  Since its first use in 1977 for the treatment of strabismus in children, BoNT-A has since been used in aesthetic medicine and for the treatment of a number of disorders associated with overactive striated muscles, such as strabismus, esotropia, exotropia , focal dystonia, spasticity, and movement disorders.
  BoNT-A has also been used in the management of some smooth-muscle disorders, such as achalasia, oesophageal spasm , ptyalism, hyperhidrosis, and intrinsic rhinitis, blepharospasm, muscle spasms and spasticity, axillary hyperhidrosis, and neurogenic detrusor muscle overactivity of the urinary bladder.
Diagnostic Test: Penile duplex and shear wave elastosonography (SWE). — Penile duplex study using intracavernosal injection of prostaglandin E1 (PGE1) before and after Botox injection (in the follow-up visit in the 6th week after Botox injection). Penile cavernosal arteries diameters and colored waves will be assessed. Shear wave elastosonography will be conducted comparing the stiffness of penile tissues before and after Botox injection

SUMMARY:
The goal of this clinical trial is to find out if injecting Botox into men with erectile dysfunction makes their penis less stiff and gives them better erections. This will be done using a new ultrasound method. The main questions it tries to answer are: Is Botox injection safe and effective for men suffering from erectile dysfunction who failed other treatment methods? Does this new method have any radiological criteria for penile tissues? • If Botox is injected into the penis, is there a cut-off number for this technique that shows how much better things are before and after? Before and after treatment, participants will rate how much their erections have improved, and investigators will connect their answers to the findings

ELIGIBILITY:
Inclusion Criteria:

* Men with ED not responding to oral PDE5Is.

Exclusion Criteria:

* Patients with penile prostheses.
* Patients diagnosed with Peyronie's disease.
* Non-vascular erectile dysfunction.
* Medical comorbidities that would limit the benefit of ICI such as uncontrolled diabetes mellitus, significant cardiovascular disease interfering with sexual activity, unstable psychiatric conditions, and the presence of anatomical, hormonal, or neurological abnormalities that would significantly impair erectile function.
* Patients with a history of radical pelvic surgery.
* Pelvic or spinal trauma

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
The International Index of Erectile Function Questionnaire (IIEF-5) score in patients with erectile dysfunction correlated with penile elasticity. | 1 months
  The International Index of Erectile Function Questionnaire (IIEF-5) is a questionnaire used by patients suffering from Erectile dysfunction to subjectively grade their condition. The score range from 5-25. and the erection status is classified into five categories based on the score: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), no erectile dysfunction (22-25). The higher the score, the better the erection state.
Change from baseline in penile hardness using Shear wave elastosonography (SWE) after Intracavernosal injection by Botox at 6 weeks. | 6 weeks
  An elastosonographic method was introduced as a new ultrasound technique that provides information regarding the rigidity of tissues rather than their morphology. There are two types of elastosonographic methods: strain elastosonography and shear wave elastosonography (SWE). The unit used is kilopascals. The lower the values, the better the outcome. Rigid penis has stiffer tissues which have lower SWE values.
Change from baseline in the IIEF-5 score after Intracavernosal injection by Botox at 6 weeks. | 6 weeks
  The International Index of Erectile Function Questionnaire (IIEF-5) is a questionnaire used by patients suffering from Erectile dysfunction to subjectively grade their condition. The score range from 5-25. and the erection status is classified into five categories based on the score: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), no erectile dysfunction (22-25).

SECONDARY OUTCOMES:
A cut-off SWE value for determining significant pathological degree of elasticity of the cavernous tissue that would possibly benefit from ICI treatment by Botox | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No